CLINICAL TRIAL: NCT07141641
Title: Individual Patient Expanded Access for Acellular Tissue Engineered Vessel (ATEV) for Vascular Disease and Dialysis Access
Status: Temporarily not available | Type: Expanded Access
Sponsor: Humacyte, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CLN-EA-IP-2
Record Dates: First submitted 2025-08-19; First posted 2025-08-26 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-08

CONDITIONS: Vascular Diseases; End Stage Renal Disease on Dialysis
MeSH Terms: conditions — Vascular Diseases

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Biological: Acellular Tissue Engineered Vessel (ATEV)

SUMMARY:
Individual patient expanded access requests may be considered for patients who have no other treatment options and are not eligible for an ATEV clinical study.

DETAILED DESCRIPTION:
Procedure for Requesting Expanded Access:

The treating physician requesting expanded access must contact Humacyte directly with the basis for the request. Please include the Investigator's contact information so that Humacyte may follow up with the Investigator directly.

General Criteria:

The Humacyte Expanded Access Committee will evaluate and respond to each expanded-access request received on a case-by-case basis. Humacyte will consider the nature of the request, the patient's health, the available medical and scientific information about the investigational product, the balance of risk and potential benefit to the patient, the availability of investigational product, and the potential regulatory impact.

Anticipated Timing:

Humacyte will acknowledgement receipt of each Investigator request within ten (10) business days or less.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

-

Age Groups: Child, Adult, Older Adult